Effect mechanism of custom-made foot orthoses on foot pronation subjects and

chronic low back pain: a randomized controlled trial

Study Design: Double blinded Randomized controlled trial.

Clinical Relevance

Custom-made foot orthoses may contribute to improving chronic low back pain. This

question represents an important benefit for patients and for the public health system by

reducing expensive treatments, such as surgery or long periods of rehabilitation.

Keywords Low back pain, foot, pronation, posture, custom-made foot orthoses.

NCT number NCT03996980

Date: 4/02/2019

Methods

Design

A double-blinded two-arm randomized controlled trial. The participants were randomly

allocated to a custom-made foot orthoses intervention group or a placebo orthoses

intervention group.

This paper was written according to the CONSORT 2010 Statement guideline for

reporting randomized clinical trials (Schulz KF, Altman DG, Moher D, CONSORT

Group.

# Recruitment

The trial was conducted between January 2019 and September 2019. The participants were between 18 and 65 years old with a diagnosis of nonspecific CLBP and pronated foot (FPI  $\geq$  +6) recruited from the Podiatry Clinic of the University of Seville. Potential participants were initially interviewed briefly to be evaluated in the participation in the study (a qualified podiatrist carried out this initial assessment). The original sample consisted of 105 subjects (54 women and 51 men), 53 corresponding to the experimental group and 52 to the control group. After finishing the follow-up period, there was a loss of 4 subjects (who left the study for unknown reasons or because it was impossible to contact them).

# Inclusion Criteria

The inclusion criteria were: Males and females between 18 and 65 years old, presence of CLBP, Foot Posture Index pronated in one or both feet (henceforth, FPI)  $\geq +6^{16}$ .

# **Exclusion Criteria**

The exclusion criteria were: serious illness, current participation in another research study, pregnancy, previous back or foot surgery, current treatment of foot pathology or back, and leg length discrepancy > 5 mm

### Procedure

We recruited 105 patients of the Podiatry Area of the University of Seville. There was a routine biomechanical lower limb examination to determine the inclusion criteria (Figure 1). A <u>podiatrist</u> assessed the foot posture during the biomechanical assessment based on the six-item foot posture index (FPI≥+6) <sup>16</sup>. The FPI consists of six validated

items measured in a standing relaxed position of the subject; The categories are:

Supinated foot: -1 a -12.

Neutral foot posture: 0 to +5 (neutral).

Pronated foot posture: +6 to +12.

The patients were randomized to either an experimental treatment group or a control

group. The main researcher and the participants were blind to which group and kind of

treatment was being studied. The random allocation to each group was done by a

collaborating researcher who generated the random sequence ( blocked randomization

based on a random numbers table) and the treatment was administered

(experimental/control).

The primary outcome was measured at the moment of inclusion in the study, and after

four weeks of use of the orthose treatment. We used the Oswestry Disability Index

Questionnaire (ODI) for Lower Back Pain which provides information on disability due

to CLBP and its impact on ten daily activities and a 100 mm visual analogue scale (VAS).

At the end of the study the control group received the custom-made foot orthoses best

suited to them.

Fabrication of foot orthoses

Molds of both feet were obtained for all the participants. The phenolic foam molds were

made in a condition of the participant's feet under weight-bearing. The feet were

manipulated before being introduced into the phenolic foam placed in a neutral position.

We obtained a positive mold of the feet filling the phenolic foam molds with liquid plaster.

The positive mold was used to make the custom orthoses of polypropylene of 3-

mm (heated to 180°C) from the heel to just behind the metatarsal heads, covered with a 2-mm thick polyethylene foam layer of 35-shore in the experimental group. For the control group, placebo treatment, a flat insole was made of polyester resin adjusting it to the size of the foot, but not adapting it, the aim being not to alter the patient's normal function (Figure 1).



Figure 1. Foot orthoses.

# Statistical analysis

The recruitment target was 101 participants (G\* Power 3.0.10, Franz Faul, Universität Kiel, Germany). Based on a preliminary study<sup>12</sup> the sampling size necessary was 36 participants in each group. This size was increased to compensate for possible alterations in the statistical significance of the results caused by potential participant dropouts. Therefore, we used a final sample size of a total of 101 participants.

The Student's t test was used for the comparison between means and medians of the groups. Whenever a normally distribution pattern was rejected, the nonparametric Mann–Whitney U test was applied. Secondary outcomes were tested for differences by Pearson's Chi² or Student's t-tests.

All analyses were performed using SPSS® version 24.0. A P-value <0.05 was set as statistically significant.



# **REFERENCES** 1. Chuter V, Spink M, Searle A. The effectiveness of shoe insoles for the prevention and treatment of low back pain: a systematic review and metaanalysis of randomised controlled trials. BMC Musculoskelet Disord 2014); 15 (1): 140-8.

- 2 Kendall, J, Bird, AR, Azari, MF Foot posture, leg length discrepancy and low back pain-Their relationship and clinical management using foot orthoses- An overview. Foot 2014; 24(2):75-80.
- 3 Prasad A, Choudhury D. Association between hyper-pronated foot and the degree of severity of disability in patients with non-specific low back pain. J of bodyw mov ther 2018; 22: 757-60.
- 4 Farahpour N, Jafarnezhadgero A, Allard P, Majlesi M. Muscle activity and kinetics of lower limbs during walking in pronated feet individuals with and without low back pain. J Biomech 2018; 39: 35-41.
- 5.Ferrari R. Responsiveness of the short-form 36 and Oswestry disability questionnaire in chronic nonspecific low back and lower limb pain treated with customized foot orthotics. J Manipulative Physiol Ther 2007; 30(6):456-8.
- 6 Brantingham, JW, Lee Gilbert, J, Sheik, J., Globe, G. Sagittal plane blockage of the foot, ankle and hallux and foot alignment-prevalence and association with low back pain, Journal of Chiropractic Medicine 2006;5(4);123-7.
- 7 Pinto, RZ, Souza T.R., Trede RG, Kirkwood R.N., Figueiredo, E.M., Fonseca, S.T. Bilateral and unilateral increases in calcaneal eversion affect pelvic alignment in standing position. Man Ther 2008; 13(6):513-519.
- 8 Cambron, J.A., Duarte, M., Dexheimer, J., Solecki T. Shoe orthotics for the treatment of chronic low back pain: a randomized controlled pilot study. J Manipulative Physiol Ther 2011; 34(4):254-260.
- 9 Farokmanesh K., Shirzadian T., Mahboubi M., Neyakan M. Effect of foot hyperpronation on lumbar lordosis and thoracic kyphosis in standing position using 3-dimensional ultrasound-based motion analysis system. Glob J Health Sci 2014; 6 (5): 254-9.

- 10 O'Leary C., Cahill C., Robinson A., Barnes M., Hong H. A systematic review: the effects of podiatrical deviations on nonspecific chronic low back pain. J Back Musculoskelet Rehabil 2013;26(2): 117-23.
- 11 Livingnstone L.A., Mandingo J.L. Bilateral rear foot asymmetry and anterior knee pain syndrome. J Orthop Deportes Phys Ther 2003; 33(1):48-54.
- 12 Castro-Méndez, A., Munuera, P.V., Albornoz-Cabello,M. The short-term effect of custom-made foot orthoses in subjects with excessive foot pronation and lower back pain: A randomized, double-blinded, clinical trial. Prosthetics and Orthotics 2012; 37(5); 384-390.
- 13 Papúa,M.O., Cambron,J. Foot orthotics for low back pain: the state of our understanding and recommendations for future research. Foot 2016. 26:53-7.
- 14 Rosner A, Conable K, Eldelmann T. Influence of foot orthotics upon duration of effects of spinal manipulation in chronic back pain patients: A randomized clinical trial. J Manipulative Physiol Ther 2013; 37 (2):124-40.
- 15 Zahran S., Ale S., Zaky L. Effects of bilateral flexible flatfoot on trunk and hip muscles'torque. Rehabilitación Int J Ther 2017; 24(1):7-14.
- 16. Pascual Gutierrez R, Redmon AC, Alcacer Pitarch B, López Ros P. Índice de postura del pie (IPP-6), versión de seis criterios. Manual y guía de usario. Podología clínica 2013; 14(2):36-45.
- 17 Ghasemi M., Koohpayehzadeh J, Kadkhodaei H., Ehsani A. The effect of foot hyperpronation on spine alignment in standing position. MJIRI 2016;30:466-72.
- 18 Resende R.A, Kirkwood R.N., Deluzio K.J., Fonseca T.S. Ipsilateral and contralateral foot pronation affect lower limb and trunk biomechanics of individuals with knee osteoarthritis during gait. Clin Biomech 2016; 7:30-7.

- 19. Resende A., Deluzio K., Kirkwood R, Hassan A., Fonseca, S. Increased unilateral foot pronation affects lower limbs and pelvic biomechanics during walking. Gait & Posture 2015; 41(2):395-401.
- 20.Sahar T, Cohen MJ, Uval-Neeman V, Kandel L, Odebiyi DO, Lev I, et al. Insoles for prevention and treatment of back pain: a systematic review within the framework of the Cochrane Collaboration Back Review Group. Spine 2009; 34(9):924-933.
- 21. Dananberg, H.J. Sagittal plane biomechanics. J AM Podiatr Med Assoc 2000; 90(1):47-50.
- 22. Khamis S., Yizhar Z. Effect of feet hyperpronation on pelvic alignment in a standing position. Gait Posture 2007; 25(1):127-134.
- 23. Declaración de Helsinki de la AMM Principios éticos para las investigaciones médicas en seres humanos. Asamblea General de la AMM, Fortaleza, Brazil, October 2013.
- 24. Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP. Declaración de la Iniciativa STROBE (Strengthening the Reporting of Observational studies in Epidemiology): directrices para la comunicación de estudios observacionales. Gac Sanit. 2008; 22(2):144-50.
- 25 Knutson G.A. Anatomic and functional leg-length inequality: a review and recommendation for clinical decision-making. Part I, anatomic leg-length inequality: prevalence, magnitude, effects and clinical significance. Chiropr Osteopat. 2005;20;11-3.
- 26 Alcántara-Bumbiedro S., Flórez-García M.T., Echávarri-Pérez C., García-Pérez F. Escala de incapacidad por dolor lumbar de Oswestry. Rehabilitación: Revista de la Sociedad Española de Rehabilitación y Medicina Física. 2006;40;

- 3:150-158.
- 27 Bijur P., Silver W., Gallagher E. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med 2001; 8(12):1153-1157.
- 28 Yazdani S. Dizji E., Alizadeh F, Hassanlouei H. Effect of chronic idiopathic low back pain on the kinetic gait characteristics in different foot masks. J Biomech 2018; 79:243-7.
- 28. Kelvin J., Molyneux T., Le Grande M., Castro A., Franz K., Fuss, M.D., Azari M. Association of Mild Leg Length Discrepancy and Degenerative Changes in the Hip Joint and Lumbar Spine. JMPT 2017;40(5):301-9.
- 29.Kim S.C., Yi J.H., Jung S.W., Seo D.K. The effects of calcaneal posture on thoracolumbar alignment in a standing position. J Phys Ther Sci. 2017;29(11):1993-5.